CLINICAL TRIAL: NCT03627559
Title: Early Detection of Anastomotic Leakage by Microdialysis Catheters: An Observational Study on Pancreaticoduodenectomy
Brief Title: Early Detection of Anastomotic Leakage by Microdialysis Catheters
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Espen Lindholm, senior Researcher, Oslo University Hospital
Other Study IDs: 2012/143
Record Dates: First submitted 2018-07-09; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Pancreatic Cancer; Pancreaticoduodenal; Fistula; Pancreas; Fistula; Pancreatic Fistula
Keywords: Pancreaticoduodenectomy; Pancreatectomy
MeSH Terms: conditions — Pancreatic Neoplasms; Fistula; Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Microdialysate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreaticoduodenectomy patients: All patients undergoing pancreaticoduodenectomy receive a microdialysis catheter before skin closure and will be monitored postoperatively for lactate, pyruvate, glucose and glycerol in the microdialysate at certain timepoints
  Interventions: Procedure: Pancreaticoduodenectomy microdialysis catheter analyses

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy microdialysis catheter analyses — A thin microdialysis catheter is implanted before skin closure after pancreaticoduodenectomy. Analyses of the microdialysate are done at certain timepoints postoperatively. No intervention is done based on the results. The patients are following standard of care.

SUMMARY:
Anastomotic leakage of the pancreatojejunostomy is often discovered with considerable delay, causing severe peritonitis, hemorrhage due to erosion of vessels, sepsis, and death. Microdialysis catheters can detect focal inflammation and ischemia, and has a potential for early detection of anastomotic leakage. This observational study will examine if monitoring with microdialysis catheters can detect anastomotic leakage after pancreaticoduodenectomy earlier than current standard of care.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (Whipple´s procedure) offers the only potential cure for patients with tumor in the head of the pancreas, bile duct or periampullary region. This procedure is associated with high perioperative and postoperative mortality and morbidity. Postoperative pancreatic fistulae (POPF) is the most feared complication, and is often discovered with significant delay resulting in development of organ dysfunction and sepsis. Current standard for clinical detection of POPF is limited and nonspecific.

Microdialysis catheters allow bedside measurements of metabolism such as lactate, pyruvate, glucose and glycerol. The method has a high sensitivity and specificity in detecting complications in several types of abdominal surgery. However, microdialysis used after pancreaticoduodenectomy is not well documented. This observational study examine if monitoring with microdialysis catheters can detect anastomotic leakage after pancreaticoduodenectomy earlier than current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Tumor in the head of the pancreas, the bile duct or the duodenum detected on a computed tomography (CT) scan or magnetic resonance imaging (MRI), and evaluated by a multidisciplinary team to be resectable with a pancreaticoduodenectomy.
* Written informed consent was obtained before study enrollment.

Exclusion Criteria:

* <18 years
* patient with tumor which was not resectable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both genders from age 18 and older. Tumor in the head of the pancreas, the bile duct or the duodenum. Planned to undergo pancreaticoduodencetomy
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Glycerol concentration postoperatively | Measured hourly during the first 24 hours and thereafter every 2-4 hours during hospitalization at an average of 10 days after surgery
  Glycerol concentration of the microdialysate is measured hourly during the first 24 hours and thereafter every 2-4 hours during hospitalization at an average of 10 days after surgery
Glucose concentration postoperatively | Measured hourly after surgery during the first 24 hours and thereafter every 2-4 hours during hospitalization at an average of 10 days after surgery
  Glucose concentration of the microdialysate is measured hourly during the first 24 hours and thereafter every 2-4 hours during hospitalization at an average of 10 days after surgery
Lactate concentration postoperatively | Measured hourly after surgery during the first 24 hours after surgery and thereafter every 2-4 hours during hospitalization at an average of 10 days after surgery
  Lactate concentration of the microdialysate is measured hourly during the first 24 hours and thereafter every 2-4 hours during hospitalization at an average of 10 days after surgery
Pyruvate concentration postoperatively | Measured hourly after surgery during the first 24 hours and thereafter every 2-4 hours during hospitalization at an average of 10 days after surgery
  Pyruvate concentration of the microdialysate is measured hourly during the first 24 hours and thereafter every 2-4 hours during hospitalization at an average of 10 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Espen Lindholm, ph.d, Principal Investigator — Oslo University Hospital

IPD SHARING:
Plan to Share IPD: No
No plan for share IPD

REFERENCES:
- [Derived] Lindholm E, Bergmann GB, Haugaa H, Labori KJ, Yaqub S, Bjornbeth BA, Line PD, Grindheim G, Kjosen G, Pischke SE, Tonnessen TI. Early detection of anastomotic leakage after pancreatoduodenectomy with microdialysis catheters: an observational Study. HPB (Oxford). 2022 Jun;24(6):901-909. doi: 10.1016/j.hpb.2021.10.020. Epub 2021 Nov 5. PMID 34836755